CLINICAL TRIAL: NCT00370110
Title: A Double-blind, Randomized, Placebo-controlled, Single Center, Parallel Group Study to Evaluate the Effects of Itopride (100 mg and 200 mg t.i.d.) on Gastric Motor and Sensory Functions in Healthy Volunteers
Brief Title: Effects of Itopride on Gastric Motor and Sensory Functions in Healthy Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITODG04-02
Record Dates: First submitted 2006-08-28; First posted 2006-08-30 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Healthy
MeSH Terms: interventions — itopride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Itopride (Experimental)
  Interventions: Drug: Itopride 100 mg; Drug: Itopride 200 mg
- Placebo (Other)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Itopride 100 mg — 100 mg three times daily
  Arms: Itopride
Other: Placebo
  Arms: Placebo
Drug: Itopride 200 mg — 200 mg three times daily
  Arms: Itopride

SUMMARY:
Itopride is a new compound that is already marketed in Japan and in some countries of Eastern Europe under the name of Ganaton. It is used to treat symptoms associated with gastroparesis. Due to inadequate gastric emptying, these patients often have symptoms of bloating, nausea and vomiting following ingestion of a meal. This is a randomized, parallel group, two dose double blind, placebo-controlled study evaluating the effects of itopride (100 mg and 200 mg three times daily) and placebo on gastric motor and sensory functions in healthy volunteers.

DETAILED DESCRIPTION:
In order to compare the effects of two itopride doses (100 mg and 200 mg three times daily) and placebo on gastric emptying and small bowel transit, gastric accommodation, and postprandial symptoms in female and male healthy volunteers, the following methods, which have been extensively used and validated in the laboratory, will be used:

Scintigraphic gastric emptying of solids and small bowel transit; single photon emission computed tomography to measure gastric accommodation; and the nutrient drink test to measure maximum tolerated volume and postprandial symptoms.

Based on data acquired using the same methods in the laboratory, the sample size of 15 subjects per group provides 80% power to detect an effect size of 16% in the primary endpoint of the study, that is a change in gastric volume (postprandial - fasting). This magnitude of change is considered clinically relevant.

ELIGIBILITY:
Inclusion Criteria:

1.Non-pregnant, non-breastfeeding females 2.18 years of age or older 3.Body mass index between 20 and 32 kg/m2 4.No alarm indicators on clinical assessment (weight loss of more than 7 kg, bleeding, recent recurrent vomiting, progressive dysphagia).

5.No history suggestive of small bowel obstruction

Exclusion Criteria:

1. Patients who have any gastrointestinal symptoms. Do not fulfill the criteria for the irritable bowel syndrome or functional dyspepsia clinically
2. Patients with a clinical diagnosis of gastroparesis or an alternative underlying disease that could be responsible for disturbed gastric function e.g. diabetes, post-vagotomy, post-fundoplication
3. Abdominal surgery other than appendectomy, cholecystectomy, hysterectomy, caesarian section or tubal ligation
4. Positive symptoms on an abridged bowel disease questionnaire
5. Use of medications that may alter gastrointestinal motility including metoclopramide, domperidone, tegaserod; acetaminophen and ibuprofen will be allowed
6. Current use of medications which may interact with the study medications
7. Patients who have taken any investigational medications within the past 30 days
8. Over the counter medication (except multivitamins) within 7 days of the study
9. Chronic gastrointestinal illness or any systemic disease that could affect gastrointestinal motility for controls
10. Known intolerance or allergy to eggs, milk and Ensure
11. History of chronic diarrhea

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-08; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Gastric emptying | one week

SECONDARY OUTCOMES:
Small bowel transit | one week
Gastric accommodation | one week
Postprandial symptoms | one week

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J. Talley, M.D., Ph.D., Principal Investigator — Mayo Clinic College of Medicine
Locations (1):
- Mayo Clinic College of Medicine, Rochester, Minnesota, United States